Effect of health education by feedback method on postoperative rehabilitation and compliance behavior of patients with lumbar disc herniation

(February 25, 2019)

## **Appendix**

# Appendix 1: Informed Consent Form

#### Medical Ethics Review Form

Application date: February 25, 2019

**Project Name:**Effect of health education by feedback method on postoperative rehabilitation and compliance behavior of patients with lumbar disc herniation

Ethical Number: 2019082.

Project Leader: Fan Rong

Research team members: Fan Rong, Fan LiAng, Zhang Min

Research Project Source: Tianjin Hospital Department Project

Submission of Examination Information: 

□plan □Informed consent

### A summary of biomedical research contents and research protocols involving humans

Based on feedback method, health education for postoperative rehabilitation compliance behavior of patients with lumbar disc herniation was constructed Plan; Comparing this plan with conventional care in disease knowledge, compliance behavior and patients with lumbar disc herniation Functional recovery and other aspects of the difference. Make clear that this feedback method of health education program in improving the patient's knowledge of water The application value of smoothing, complying with medical behavior and improving postoperative lumbar function is further improved and developed. The intervention methods for such patients provide reference basis.

### Review opinions of the ethics committee of the unit

After the discussion by the medical ethics committee of Tianjin hospital, the design of the experimental scheme is reasonable and it can be guaranteed well Subject rights, the investigator is qualified to participate in the clinical trial. Agreed to carry out the experiment.

Chapter of the Medical Ethics Committee:

February 25, 2019

# Appendix 2

(1) Explanation of the knowledge of the experimental group and watching the intraoperative video.









(2) The control group received routine health education.



(3) The experimental group was given functional exercise feedback.



# Appendix 3 Post-discharge health education

- 1. The patients in the experimental group were given knowledge feedback, and the patients needed to give specific knowledge points in their own language.
- 2. The experimental group received feedback of functional exercise in the form of video.



- 3. The convalesives were invited to make comments and corrections on the functional exercise methods of the patients, and the researchers would feedback the comments to the patients.
- 4. WeChat answers questions from patients at any time.
- 5.Outpatient review: questionnaires were completed and functional exercise responses were given, such as walking training and straight leg raising exercises.



6.The control group received the explanation of knowledge and functional exercise, and only needed to reply and receive.